CLINICAL TRIAL: NCT04850339
Title: A Randomized, Double-Blind, Placebo-Controlled, Ascending Single and Multiple Dose First in Human Study to Evaluate the Safety, Tolerability and Pharmacokinetics of ANXV Administered as an Intravenous Infusion to Healthy Male Subjects
Brief Title: First in Human Study of ANXV (Recombinant Human Annexin A5) in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Annexin Pharmaceuticals AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ANN-001
Record Dates: First submitted 2021-03-04; First posted 2021-04-20 (Actual); Last update posted 2022-05-16 (Actual); Status verified 2022-05

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- ANXV single dose (Active Comparator): ANXV in a single ascending dose pattern in four dose levels.
  Interventions: Biological: ANXV
- Placebo single dose (Placebo Comparator): Placebo in a single ascending dose pattern in four dose levels.
  Interventions: Other: Placebo
- ANXV multiple dose (Active Comparator): ANXV in a multiple ascending dose pattern in three dose levels.
  Interventions: Biological: ANXV
- Placebo multiple dose (Placebo Comparator): Placebo in a multiple ascending dose pattern in four dose levels.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: ANXV — Intravenous infusion
  Arms: ANXV multiple dose; ANXV single dose
Other: Placebo — Intravenous infusion
  Arms: Placebo multiple dose; Placebo single dose

SUMMARY:
This is an adaptive, randomised, double-blind, single-centre, placebo-controlled phase I, First in Human study designed to evaluate the safety, tolerability and pharmacokinetics of single and multiple intravenous dosing of ANXV in healthy male subjects.

DETAILED DESCRIPTION:
This First in Human study is divided in two parts. Part I, Single Ascending Dose (SAD), will explore safety, tolerability and PK of single intravenous doses of ANXV. Part II, Multiple Ascending Dose (MAD), will explore safety, tolerability and PK of multiple doses (five consecutive daily doses) of intravenous ANXV.

The objectives of this study are:

Primary objective:

- To evaluate the safety and tolerability of single/multiple ascending doses of ANXV in healthy male subjects.

Secondary objective:

- To determine the PK profile of single/multiple ascending doses of ANXV in healthy male subjects.

Exploratory objectives:

- To evaluate ADA to ANXV and other relevant parameters.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to give written informed consent for participation in the study.
2. Healthy male subject aged 18-50 years inclusive at screening.
3. BMI ≥ 18.0 and ≤ 30.0 kg/m2 and weight at least 50 kg and no more than 100 kg at screening.
4. Overtly healthy based on medical history, physical findings, vital signs, ECG and laboratory values at the time of screening, as judged by the Investigator.
5. Male subjects must be willing to use condom or be vasectomised or practice sexual abstinence to prevent pregnancy and drug exposure of a partner, and refrain from donating sperm from the date of dosing until 3 months after (last) dosing with the IMP. Their female partner of child-bearing potential are expected to use contraceptive methods with a failure rate of < 1% to prevent pregnancy (combined [oestrogen and progestogen containing] hormonal contraception associated with inhibition of ovulation [oral, intravaginal, transdermal], progestogen-only hormonal contraception associated with inhibition of ovulation [oral, injectable, implantable], intrauterine device [IUD] or intrauterine hormone-releasing system [IUS]).

Exclusion Criteria:

1. History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study.
2. Any clinically significant illness, medical/surgical procedure or trauma within 4 weeks of the first administration of IMP.
3. Malignancy within the past 5 years with the exception of in situ removal of basal cell carcinoma.
4. Any planned major surgery within the duration of the study.
5. Any positive result on screening for serum hepatitis B surface antigen (HbsAg), hepatitis C antibody and Human Immunodeficiency Virus (HIV).
6. History of thromboembolic events.
7. History of significant bleeding (gross haematuria, haemoptysis, gastrointestinal tract bleeding).
8. Evidence or history of a hypercoagulable state (e.g. shortened APTT).
9. Prior exposure to recombinant Annexin A5 (for diagnostic purposes).
10. Any history of coronary artery disease or cerebrovascular accident.
11. Known cardiac disease, cardiac anomaly or cardiac deformity.
12. Known heredity for autoimmune disease with described presence of potentially pathogenic Annexin A5 antibodies, e.g. antiphospholipid syndrome, systemic lupus erythematosus or systemic sclerosis, as judged by the Investigator.
13. Any history of or active peptic ulcer disease.
14. Any clinically significant disease affecting the respiratory tract (e.g. obstructive and restrictive respiratory disease, chronic respiratory disease such as alveolitis, inflammatory respiratory disease, autoimmune respiratory disease, present respiratory infections, pulmonary vascular disease) that would influence the results of the study or the subject's ability to participate in the study, as judged by the Investigator.
15. eGFR (based on plasma-creatinine) outside of normal range at screening or known renal impairment (≤70 mL/min).
16. Vaccination with live-attenuated vaccines within 4 weeks of the screening visit.
17. After 5 minutes supine rest at the time of screening, any vital signs values outside the following ranges:

    * Systolic blood pressure <90 or >140 mmHg, or
    * Diastolic blood pressure <40 or >90 mmHg, or
    * Pulse <40 or >100 bpm
18. Current evidence or history of bacterial, viral or fungal infections within 7 days before (first) IMP administration as judged by the Investigator.
19. Prolonged QTcF (>450 ms), cardiac arrhythmias or any clinically significant abnormalities in the resting ECG at the time of screening, as judged by the Investigator.
20. History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the Investigator, or history of hypersensitivity to drugs with a similar chemical structure or class to ANXV.
21. Regular use of any prescribed or non-prescribed medication including antacids, analgesics, herbal remedies, vitamins and minerals within two weeks prior to the (first) administration of IMP, except occasional intake of paracetamol (maximum 2,000 mg/day; and not exceeding 3,000 mg/week), at the discretion of the Investigator and nasal decongestants without cortisone, antihistamine or anticholinergics for a maximum of 10 days, at the discretion of the Investigator.
22. Planned treatment or treatment with another investigational drug within 3 months prior to Day -1. Subjects consented and screened but not dosed in previous phase I studies are not excluded.
23. Current smokers or users of nicotine products. Smokers that stopped smoking <3 months prior to screening.
24. Positive screen for drugs of abuse or alcohol at screening or on admission to the unit prior to administration of the IMP.
25. History of alcohol abuse or excessive intake of alcohol, as judged by the Investigator.
26. Presence or history of drug abuse, as judged by the Investigator.
27. History of, or current use of, anabolic steroids.
28. Excessive caffeine consumption defined by a daily intake of >5 cups of caffeine containing beverages.
29. Intake of xanthine and/or taurine containing energy drinks within 2 days prior to screening.
30. Plasma donation within one month of screening or blood donation (or corresponding blood loss) of >450 ml during the three months prior to screening.
31. Investigator considers the subject unlikely to comply with study procedures, restrictions and requirements, or unfit for participation for any other reason.
32. Previous confirmed COVID-19 disease requiring hospital care or positive COVID-19 test on admission to the clinic.
33. Insufficient venous access for study procedures.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2020-12-21 (Actual); Primary Completion 2021-10-27 (Actual); Study Completion 2021-10-27 (Actual)

PRIMARY OUTCOMES:
Frequency of adverse events. | From day 1 (inclusion) until day 35
  Frequency of adverse events at single and multiple ascending doses of ANXV.
Seriousness of adverse events. | From day 1 (inclusion) until day 35
  Seriousness of adverse events at single and multiple ascending doses of ANXV.
Intensity of adverse events. | From day 1 (inclusion) until day 35
  Intensity of adverse events at single and multiple ascending doses of ANXV.

SECONDARY OUTCOMES:
PK profile of single and multiple ascending doses of ANXV: AUClast | 0-24hours after IMP administration
  AUC from time zero to time of last quantifiable analyte concentration (AUClast)
PK profile of single and multiple ascending doses of ANXV: Cmax | 0-24hours after IMP administration
  Observed maximum concentration (Cmax)
PK profile of single and multiple ascending doses of ANXV: Tmax | 0-24hours after IMP administration
  Time to Cmax (Tmax)
PK profile of single and multiple ascending doses of ANXV: λz | 0-24hours after IMP administration
  Terminal slope of a semi-logarithmic concentration-time curve (λz)
PK profile of single and multiple ascending doses of ANXV: T½ | 0-24hours after IMP administration
  Terminal half life (T½)
PK profile of single and multiple ascending doses of ANXV: CL | 0-24hours after IMP administration
  Clearance (CL)
PK profile of single and multiple ascending doses of ANXV: Vz | 0-24hours after IMP administration
  Volume of distribution (Vz)
PK profile of single and multiple ascending doses of ANXV: Fraction excreted in urine (fe) | 0-24hours after IMP administration
  Fraction excreted in urine (fe)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Frostegård, MD, PhD, Study Director — Annexin Pharmaceuticals
Locations (1):
- QPS Netherlands B.V., Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No